CLINICAL TRIAL: NCT04113070
Title: The Effect of Childhood Overweight and Obesity and Genetic Factors on Puberty Development: a Prospective Cohort Study
Brief Title: Overweight and Obesity and Puberty Development Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Children's Medical Center (Other); BoAi Hospital of Zhongshan (Other); QuFu People's Hospital (Individual); Inner Mongolia People's Hospital (Other)
Responsible Party: Principal Investigator, Sijia Gu, staff of Research Department, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SCMCIRB-K2019007
Record Dates: First submitted 2019-09-20; First posted 2019-10-02 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Precocious Puberty; Overweight and Obesity
Keywords: Child health care; Weight status; Environment; puberty
MeSH Terms: conditions — Puberty, Precocious; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood sample: Part of overweight and obesity and normal weight participants are required to provided venous blood sample to test their hormone level from serum fraction and analysis risk genes from plasma fraction at baseline and 1st follow-up period.
  2. Urine sample: Part of overweight and obesity and normal weight participants are required to provided urine sample to test environment endocrine disruptors exposed level at baseline and 1st follow-up period.
  3. Stool sample: Part of overweight and obesity and normal weight participants are required to provided stool sample to test their enteric microorganism at baseline and 1st follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overweight and obesity group: 1. Children with BMI cutoff points greater than 25.0 or 30.0 at 18 years old were defined overweight or obesity according to age- and sex-specific cutoff points standard proposed by International Obesity Task Force (IOTF) for 2- to 18-year-old children.
  2. Willingness to comply with study requirements
  Interventions: Device: Anthropometric measuring; Other: Growth environment evaluation
- Non-overweight group: 1. Children with BMI smaller than 25.0 at 18 years old were defined non-overweight according to age- and sex-specific cutoff points standard proposed by International Obesity Task Force (IOTF) for 2- to 18-year-old children.
  2. Willingness to comply with study requirements
  Interventions: Device: Anthropometric measuring; Other: Growth environment evaluation

INTERVENTIONS:
Device: Anthropometric measuring — To divide participants into overweight and obesity and non-overweight group according to their weight status, height (H), weight (W) and waist circumference (WC) will be measured with a uniform tool, which has been calibrated. When measuring the height, the subjects are required to take off their shoes and stand in an upright position. To measuring weight, the subjects are required to wear close-fitting clothes and bare feet. Subjects are required to take the standing position to measure waist circumference horizontally at the mid-point of line between the lower margin of the ribs and the upper margin of the ilium. All those data will be kept one decimal place. Anthropometric measuring will be taken at baseline and follow-up periods.
Other: Growth environment evaluation — The information of children' growth environment, including family environment, physical activities, dietary and sleep habits, will be collected by parent-report questionnaire at baseline and follow-up periods.

SUMMARY:
Precocious puberty and childhood overweight and obesity are important public health problems that both had adverse effects, which including psychological symptom in childhood, short final height or reproductive dysfunction in adulthood, on children's physical and psychological development.The prevalence of precocious puberty and childhood overweight and obesity are both high, and a growing body of epidemiological studies suggested that there was a close relationship of childhood overweight and obesity with puberty development, especially in girls. However, the underlying mechanism between them is unclear. Existing evidence shows that the occurrence of precocious puberty and overweight and obesity are the result of interaction of multiple factors, which consists growth environment and genetics, and many previous studies provided that more overlapping genes existed between obesity and precocious puberty patients, suggesting that common genes may result in these diseases. Therefore, based on a case control study, which will investigate the associations between obesity pleiotropic genes and early puberty, the researchers will collect information related to obesity, growth environment factors and risk genes in this study to evaluate the relationships of these related factors and precocious puberty, and to further explore whether there exists biological interaction effects of these risk factors on sexual precocity. This project has been approved by the Ethics Committee of Shanghai Children's Medical Center.

DETAILED DESCRIPTION:
1. Purpose: A prospective cohort study. The aim of this study is to investigate the effect of pediatric weight status and childhood growth environment on puberty development.
2. Participants: Participants are primary school children aged 6- to 12-year-old, and their parents must be willing to engage in this study and comply with study requirements.
3. Study Procedure: According to geographic and population distribution, about 40 schools included in this study by stratified, random clustering sampling in three cities of China, including Qufu, Zhongshan and Huhhot. Participant will accept anthropometric measuring by clinicians from the three collaborated hospitals, including BoAi Hospital of Zhongshan, QuFu People' s Hospital and Inner Mongolia People's Hospital. This study will be conducted among children of grade 1 to 3 from selected schools in 2019 and the first, secondary and third follow-up will be conducted one, two and three year later respectively.
4. Exposures: Participants with overweight or obesity will be included in overweight and obesity group at baseline.
5. Related risk factors: Childhood growth and family environmental information, including physical activity, diet habit, sleep duration, family structure and family social-economic status, will be collected by parent-reported questionnaire;
6. Outcomes measures: Participants' puberty stage will be evaluated by secondary sexual characteristics development by physician palpation.

ELIGIBILITY:
Inclusion Criteria:

* Children over 6 years old from grade 1, 2 and 3 in selected primary schools in Zhongshan, Qufu and Huhhot since 2019

Exclusion Criteria:

* Children with overweight or obesity had a history of hormone drug treatment last for 6 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A stratified random sample of children over 6 years old from grade 1 to 3 of selected primary schools in three cities in China
Sampling Method: Probability Sample
Enrollment: 14100 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of precocious puberty | 1 year
  All subjects will accept physician palpation to assess their puberty development stage according to Tanner staging method: Testicular volume will be measure by palpation and a Prader testicular meter and be graded to 1 (< 4 ml) to 5 (> 20 ml) in boys. Breast development will be graded to 1(pre-adolescent) to 5 (fully mature) in girls. Pubic hair development will be graded to 1(pre-adolescent) to 5 (fully mature) in both boys and girls. Precocious puberty will be defined as the onset age of breast development (B2) or pubic hair development (PH2) before 8 years or menarche before 10 years in girls and of PH2 or testicular enlargement (T2) before 9 years in boys. For girls with overweight or obesity, breast ultrasound will be used to discriminate glandular breast and fat tissue.

SECONDARY OUTCOMES:
Rate of early puberty | 1 year
  All subjects will accept physician palpation to assess their puberty development stage according to Tanner staging method: Testicular volume will be measure by palpation and a Prader testicular meter and be graded to 1 (< 4 ml) to 5 (> 20 ml) in boys. Breast development will be graded to 1(pre-adolescent) to 5 (fully mature) in girls. Pubic hair development will be graded to 1(pre-adolescent) to 5 (fully mature) in both boys and girls. Early puberty will be defined as children reached a certain puberty stage earlier than the median age of that stage. According to a large Chinese population-based study, the median ages for pubertal stages will be referenced. Moreover, the presence of menarche before 12 years in girls and of voice breaking before 13 years in boys will also be categorized as early puberty.

CONTACTS AND LOCATIONS:
Overall Officials: Shijian Liu, Ph.D, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen C, Zhang Y, Sun W, Chen Y, Jiang Y, Song Y, Lin Q, Zhu L, Zhu Q, Wang X, Liu S, Jiang F. Investigating the relationship between precocious puberty and obesity: a cross-sectional study in Shanghai, China. BMJ Open. 2017 Apr 11;7(4):e014004. doi: 10.1136/bmjopen-2016-014004. PMID 28400459
- [Background] Colmenares A, Gunczler P, Lanes R. Higher prevalence of obesity and overweight without an adverse metabolic profile in girls with central precocious puberty compared to girls with early puberty, regardless of GnRH analogue treatment. Int J Pediatr Endocrinol. 2014;2014(1):5. doi: 10.1186/1687-9856-2014-5. Epub 2014 Apr 17. PMID 24742263
- [Background] Wang M, Zhang Y, Lan D, Hill JW. The Efficacy of GnRHa Alone or in Combination with rhGH for the Treatment of Chinese Children with Central Precocious Puberty. Sci Rep. 2016 Apr 13;6:24259. doi: 10.1038/srep24259. PMID 27072597
- [Background] Luke B. Adverse effects of female obesity and interaction with race on reproductive potential. Fertil Steril. 2017 Apr;107(4):868-877. doi: 10.1016/j.fertnstert.2017.02.114. PMID 28366413
- [Background] Deng F, Tao FB, Liu DY, Xu YY, Hao JH, Sun Y, Su PY. Effects of growth environments and two environmental endocrine disruptors on children with idiopathic precocious puberty. Eur J Endocrinol. 2012 May;166(5):803-9. doi: 10.1530/EJE-11-0876. Epub 2012 Feb 8. PMID 22318748
- [Background] Boyne MS, Thame M, Osmond C, Fraser RA, Gabay L, Reid M, Forrester TE. Growth, body composition, and the onset of puberty: longitudinal observations in Afro-Caribbean children. J Clin Endocrinol Metab. 2010 Jul;95(7):3194-200. doi: 10.1210/jc.2010-0080. Epub 2010 Apr 28. PMID 20427487
- [Background] Biro FM, Khoury P, Morrison JA. Influence of obesity on timing of puberty. Int J Androl. 2006 Feb;29(1):272-7; discussion 286-90. doi: 10.1111/j.1365-2605.2005.00602.x. Epub 2005 Dec 20. PMID 16371114
- [Background] Kaplowitz PB. Link between body fat and the timing of puberty. Pediatrics. 2008 Feb;121 Suppl 3:S208-17. doi: 10.1542/peds.2007-1813F. PMID 18245513
- [Background] Abdel Ghany SM, Sayed AA, El-Deek SEM, ElBadre HM, Dahpy MA, Saleh MA, Sharaf El-Deen H, Mustafa MH. Obesity risk prediction among women of Upper Egypt: The impact of serum vaspin and vaspin rs2236242 gene polymorphism. Gene. 2017 Aug 30;626:140-148. doi: 10.1016/j.gene.2017.05.007. Epub 2017 May 4. PMID 28479386
- [Background] Grarup N, Moltke I, Andersen MK, Dalby M, Vitting-Seerup K, Kern T, Mahendran Y, Jorsboe E, Larsen CVL, Dahl-Petersen IK, Gilly A, Suveges D, Dedoussis G, Zeggini E, Pedersen O, Andersson R, Bjerregaard P, Jorgensen ME, Albrechtsen A, Hansen T. Loss-of-function variants in ADCY3 increase risk of obesity and type 2 diabetes. Nat Genet. 2018 Feb;50(2):172-174. doi: 10.1038/s41588-017-0022-7. Epub 2018 Jan 8. PMID 29311636
- [Background] Wasim M, Awan FR, Najam SS, Khan AR, Khan HN. Role of Leptin Deficiency, Inefficiency, and Leptin Receptors in Obesity. Biochem Genet. 2016 Oct;54(5):565-72. doi: 10.1007/s10528-016-9751-z. Epub 2016 Jun 16. PMID 27313173
- [Background] Euling SY, Selevan SG, Pescovitz OH, Skakkebaek NE. Role of environmental factors in the timing of puberty. Pediatrics. 2008 Feb;121 Suppl 3:S167-71. doi: 10.1542/peds.2007-1813C. PMID 18245510
- [Background] Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969 Jun;44(235):291-303. doi: 10.1136/adc.44.235.291. No abstract available. PMID 5785179
- [Background] Marshall WA, Tanner JM. Variations in the pattern of pubertal changes in boys. Arch Dis Child. 1970 Feb;45(239):13-23. doi: 10.1136/adc.45.239.13. PMID 5440182
- [Background] Bridges NA, Christopher JA, Hindmarsh PC, Brook CG. Sexual precocity: sex incidence and aetiology. Arch Dis Child. 1994 Feb;70(2):116-8. doi: 10.1136/adc.70.2.116. PMID 8129431
- [Background] Lebrethon MC, Bourguignon JP. Management of central isosexual precocity: diagnosis, treatment, outcome. Curr Opin Pediatr. 2000 Aug;12(4):394-9. doi: 10.1097/00008480-200008000-00020. PMID 10943823
- [Background] Klein KO. Precocious puberty: who has it? Who should be treated? J Clin Endocrinol Metab. 1999 Feb;84(2):411-4. doi: 10.1210/jcem.84.2.5533. No abstract available. PMID 10022393
- [Background] Sun Y, Tao FB, Su PY, Mai JC, Shi HJ, Han YT, Wang H, Lou XM, Han J, Liu J. National estimates of the pubertal milestones among urban and rural Chinese girls. J Adolesc Health. 2012 Sep;51(3):279-84. doi: 10.1016/j.jadohealth.2011.12.019. Epub 2012 Mar 15. PMID 22921139
- [Background] Sun Y, Tao F, Su PY; China Puberty Research Collaboration. National estimates of pubertal milestones among urban and rural Chinese boys. Ann Hum Biol. 2012 Nov-Dec;39(6):461-7. doi: 10.3109/03014460.2012.712156. Epub 2012 Aug 6. PMID 22862548
- [Background] Ong KK, Bann D, Wills AK, Ward K, Adams JE, Hardy R, Kuh D; National Survey of Health and Development Scientific and Data Collection Team. Timing of voice breaking in males associated with growth and weight gain across the life course. J Clin Endocrinol Metab. 2012 Aug;97(8):2844-52. doi: 10.1210/jc.2011-3445. Epub 2012 May 31. PMID 22654120
- [Derived] Yu T, Yu Y, Li X, Xue P, Yu X, Chen Y, Kong H, Lin C, Wang X, Mei H, Wang D, Liu S. Effects of childhood obesity and related genetic factors on precocious puberty: protocol for a multi-center prospective cohort study. BMC Pediatr. 2022 May 27;22(1):310. doi: 10.1186/s12887-022-03350-x. PMID 35624438